CLINICAL TRIAL: NCT00476411
Title: The Efficacy of HBV Vaccine Response and Prevalence of Occult HBV Infection in Isolated Anti HBc Between HIV Infected and HIV Un-infected Thai Patients
Brief Title: A Study to Test the Efficacy of the HBV Vaccine and to Look at the Prevalence of HBV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HIV-NAT 036
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis b Virus
Keywords: isolated HBc; HBV vaccine response; occult HBV in isolated antiHBC compared HIV to non HIV
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): HBV vaccine
  Interventions: Biological: HBV vaccine

INTERVENTIONS:
Biological: HBV vaccine — HBV vaccine 3 doses at month 0, 1, and 6

SUMMARY:
The prevalence of Hepatitis B core antigen in the Thai population is about 70 %, no data of isolated Hepatitis B core antigen is reported. Hepatitis B core antigen is observed in 10%-20% of individuals from low endemic areas of HBV infection. However, this prevalence of isolated antiHBc would be higher in endemic area of HBV infection. There is conflicting data of occult HBV infection in HIV infected patients. In Thailand, perinatal transmission is the main route of transmission which is different from developed countries. Therefore, isolated antiHBc in Thai people has longer duration than low prevalence regions. Moreover, HBV genotype C and B is common in this region. If the HBV vaccination could eliminate an occult HBV infection in these individuals, the liver related mortality might be reduced. The prevalence and clinical importance of isolated antiHBc in Thai have not been investigated yet. There is also limited data of HBV vaccine response in this setting.

DETAILED DESCRIPTION:
The prevalence of the Hepatitis B core antigen (anti-HBc)in the Thai population is about 70 %. No data of isolated anti-HBc is reported. Anti-HBc antigen is observed in 10%-20% of individuals from low endemic areas of HBV infection. The prevalence of isolated antiHBc antigen is expected to be higher in endemic areas of HBV infection. There is conflicting data of occult HBV infection in HIV-infected patients. In Thailand, perinatal transmission is the main route of HBV transmission, different from developed countries. Therefore, isolated anti-HBc in Thai people has longer duration than low prevalence regions. Moreover, HBV genotype C and B is common in this region. HBV genotype C is correlated with more cirrhosis and hepatoma than genotype B. A study from Taiwan demonstrated that HBV DNA > 100,000 copies/ml is correlated with cirrhosis and hepatoma. Sustained reduction of HBV replication lowers the risk of hepatoma in HBV related cirrhosis. If the HBV vaccination could eliminate an occult HBV infection in these individuals, the liver related mortality will be reduced.

The prevalence and its clinical importance of isolated anti-HBc in the Thai population has not been investigated yet. There is also limited data of HBV vaccine response in this setting.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adults followed at HIV-NAT and HIV-NAT affiliated hospitals and Un-infected HIV adults followed at chulalongkorn hospital and blood bank
* AntiHBc positive without HBsAg and antiHBs
* Written inform consent

Exclusion Criteria:

* Patients receiving, or with an anticipated need to receive, any concomitant medications with the potential to decrease the response to HBV vaccine such as long term steroid user, chemotherapy, cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
HBV DNA in HIV-infected patients presenting with a serological pattern of isolated anti-HBcAg compare to non HIV patients with isolated antiHBc | 1 year

SECONDARY OUTCOMES:
antiHBs titer after 2 month of third dose of HBV vaccine in both 2 groups | 1 year
liver function test after HAART in HIV patients compare between negative and positive HBV DNA | 1 year
3TC resistant after 3TC containing HAART in HIV patients with detectable HBV DNA prior treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, Principal Investigator — HIV-NAT, Thai Red Cross AIDS Research Center
Locations (1):
- HIV-NAT Thai Red Cross AIDS Research Center, Bangkok, Thailand

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org